CLINICAL TRIAL: NCT06886100
Title: Melanin Recurrence, Pain Perception and Wound Healing in Scalpel and LASER Gingival Depigmentation in Thin and Thick Phenotypes: a Comparative Clinical Study.
Brief Title: Melanin Recurrence in Scalpel and LASER Gingival Depigmentation in Thin and Thick Phenotypes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thamar University (Other)
Responsible Party: Principal Investigator, Wadhah Abdulnasser Noman Alhajj, Associate Professor Wadhah Alhajj, Thamar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: reference number (2024/4)
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Melanin Hyperpigmentation
Keywords: Depigmentation; Healing; Laser; Melanin; Pain; Phenotype
MeSH Terms: conditions — Vitiligo; Pain | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Thirty patients (60 sites) were included in this study. They had bilateral physiologic melanin hyperpigmentation in the upper anterior segment with severe grade II melanin hyperpigmentation. The patients were divided into two groups: each with fifteen patients with severe grade II melanin pigmentation, one with thin gingiva and another with thick gingiva. Melanin depigmentation was done in one side using scalpel no. 15 and other side with diode laser.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with thin gingival phenotype (Active Comparator): Thin gingival phenotypes are delicate, highly scalloped and translucent in appearance (Fig. 3). The soft tissue appears delicate and friable with a minimal amount of the attached gingiva.
  Interventions: Device: Diode laser; Device: Scalpel No 15
- Patients with thick gingival phenotype (Active Comparator): . The thick biotype is dense and fibrotic with a wide zone of attachment, thus making it more resistant to recession. Thin gingival biotype is a delicate, highly scalloped soft tissue and is more prone to recession, bleeding, and inflammation.
  Interventions: Device: Diode laser; Device: Scalpel No 15

INTERVENTIONS:
Device: Diode laser — Diode Laser is a semiconductor device similar to a light-emitting diode in which a diode pumped directly with electrical current can create lasing conditions at the diode's junction. It is used in periodontal surgery as melanin depigmentation
Device: Scalpel No 15 — The No.15 blade has a small curved cutting edge and is the most popular blade shape ideal for making short and precise incisions.

SUMMARY:
This study aimed to compare melanin pigmentation recurrence, pain perception and wound healing between laser and scalpel surgeries in thin and thick gingival phenotypes.Thirty patients (60 sites) were included in this study. They had bilateral physiologic melanin hyperpigmentation in the upper anterior segment with severe grade II melanin hyperpigmentation. The patients were divided into two groups: each with fifteen patients with severe grade II melanin pigmentation, one with thin gingiva and another with thick gingiva. Melanin depigmentation was done in one side using scalpel no. 15 and other side with diode laser.

DETAILED DESCRIPTION:
Background: Removal of unsightly pigmented gingiva is the need for a pleasant and confident smile. Many studies were done to study the melanin recurrence in both surgical and laser melanin depigmentation. To best of our knowledge, there is no published article regarding comparison of melanin recurrence between both techniques taking in consideration the gingival phenotype. So this study aimed to compare melanin pigmentation recurrence, pain perception and wound healing between laser and scalpel surgeries in thin and thick gingival phenotypes.

Methods: Thirty patients (60 sites) were included in this study. They had bilateral physiologic melanin hyperpigmentation in the upper anterior segment with severe grade II melanin hyperpigmentation. The patients were divided into two groups: each with fifteen patients with severe grade II melanin pigmentation, one with thin gingiva and another with thick gingiva. Melanin depigmentation was done in one side using scalpel no. 15 and other side with diode laser.

ELIGIBILITY:
Inclusion Criteria:

(i) Be aged at least 20 years, (ii) had bilateral physiologic melanin hyperpigmentation of gingiva (dark gums) in the anterior segment with severe grade II melanin hyperpigmentation (according to modification of melanin index categories 1977), (iii) periodontally healthy with good oral hygiene, (iv) had esthetic concern, (v) systemically healthy, (vi) no dental crowding and (vii) those willing to undergo minor surgical procedures.

Exclusion Criteria:

(i) any systemic disease associated with pathological hyperpigmentation), (ii) non-treated periodontal disease, (iii) chronic smokers, (iv) subjects with a mouth breathing habit (ii) subjects with crown restorations or fillings involving the incisal edge on anterior maxillary teeth, (v) non-compliant patients (vi) missing any of the six maxillary anterior teeth and having Millers Class III or Class IV recession (vii) pregnant or lactating females and (viii) (ix) gingival pigmentation of hemoglobin, melanoid, melanoma and carotene , (x) Gingival pigmentation adjacent to amalgam restoration, and (xi) Long-term usage of antimalarial drugs and minocycline.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Melanin recurrence | One week, three months, and six months postoperatively
  It is the reappearance of melanin pigmentation following a period of time after depigmentation.

SECONDARY OUTCOMES:
Wound healing | One week and one month after surgery.
  Wound healing was evaluated as per the list of clinical observations and patient responses as: Complete epithelization, incomplete epithelization, ulcer or tissue defect or necrosis.
Pain perception (VAS) | Immediately after surgery, one day, one week and one month postoperatively
  Pain perception via the Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be' (Fig. 1) [1]. The patient is asked to mark his pain level on the line between the two endpoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Wadhah dental center, Sanaa, Sanaa Governorate, Yemen

IPD SHARING:
Plan to Share IPD: Undecided
Because I do not understand exactly what do you mean by sharing individual participant data (IPD)

REFERENCES:
- [Background] Grover HS, Dadlani H, Bhardwaj A, Yadav A, Lal S. Evaluation of patient response and recurrence of pigmentation following gingival depigmentation using laser and scalpel technique: A clinical study. J Indian Soc Periodontol. 2014 Sep;18(5):586-92. doi: 10.4103/0972-124X.142450. PMID 25425820
- See also: It represent the site for a research which was a main source of study. — https://pubmed.ncbi.nlm.nih.gov/25425820/